CLINICAL TRIAL: NCT02256514
Title: Open Label Trial of Hepcortespenlisimut-L (V5) Immunotherapy for HCC
Brief Title: Open Label Trial of Immunotherapy for Advanced Liver Cancer
Acronym: HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Immunitor LLC (Industry)
Collaborators: Immunitor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMV5; IMMV5 (Other: Immunitor LLC)
Record Dates: First submitted 2014-09-24; First posted 2014-10-03 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: HCC; Liver Cirrhosis
Keywords: therapeutic vaccine
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daily oral dose of hepcortespenlisimut-L (Experimental): Hepcortespenlisimut-L (V5) (850 mg pill) to be administered once per day for the duration of study
  Interventions: Biological: Daily oral dose of hepcortespenlisimut-L

INTERVENTIONS:
Biological: Daily oral dose of hepcortespenlisimut-L — Oral therapeutic vaccine, hepcortespenlisimut-L (V5) to be given once-per-day with monthly check-up
  Other Names: V5

SUMMARY:
The purpose of this study is to evaluate daily dosing of oral immunotherapy hepcortespenlisimut-L (V5) in patients with advanced stage of HCC not amenable to surgical intervention or with recurrent tumor after surgery.

DETAILED DESCRIPTION:
Hepcortespenlisimut-L (V5) immunotherapy of HCC in an open label setting with baseline alphafetoprotein serum levels and CT scan image as primary endpoints with monthly follow-up thereafter. Additional endpoints will include blood biochemistry indices and safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years old and are willing and capable of providing informed consent. Both men and non-pregnant women will be included.
* HCC diagnosis documented prior to Study Entry by either cytology/histology, CT scan, and AFP serum test higher or equal to 30 IU/ml.
* All subjects with reproductive potential are advised to utilize effective contraception throughout the course of this study.
* Health score status at baseline.
* Agreement to participate in the study and to give at least 3 samples of blood for lab tests.
* Readily available home or o other address where patient can be found.

Exclusion Criteria:

* Subjects who might have already taken V5 in prior trials and have no baseline data.
* Those who met inclusion criteria can be retrospectively enrolled.
* Pregnant or breast-feeding women are excluded.
* Subjects who have taken other immunomodulatory therapies within 2 months prior to Entry: systemic corticosteroids, immune globulin (IV gamma globulin, IVIG), interferons, interleukins, pentoxifylline (Trental), thalidomide, filgrastim (G-CSF), sargramostim (GM-CSF); dinitrochlorobenzene (DNCB), thymosin alpha 1 (thymosin alpha), thymopentin, inosiplex (Isoprinosine), polyribonucleoside (Ampligen), ditiocarb sodium (Imuthiol), any locally available immune modulators, and any other therapeutic or preventive HCC vaccine.
* Subjects requiring concurrent participation in another experimental research treatment study, or who received an experimental agent within four weeks prior to Study Entry.
* Evidence of active or acute cardiac disease, epilepsy, or life-threatening diseases unrelated to HCC.
* Medical conditions such as active alcohol or substance abuse, or psychological issues that in the opinion of the local investigator would interfere with adherence to the requirements of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Effect of hepcortespenlisimut-L (V5) immunotherapy on serum levels of AFP (IU/ml) compared to baseline | minimum 3 months
  monthly check-up of AFP serum levels
Effect of hepcortespenlisimut-L (V5) immunotherapy on tumor size or clearance | minimum 3 months
  Comparison of abdominal CT scans at baseline and 3 months later

SECONDARY OUTCOMES:
Effect of hepcortespenlisimut-L (V5) immunotherapy in patients with advanced HCC on blood biochemistry parameters | 3 months
  Monthly blood biochemistry including liver function tests
Effect of hepcortespenlisimut-L (V5) immunotherapy on patients' performance | 3 months
  Monthly evaluation of clinical symptoms as per ECOG performance status

CONTACTS AND LOCATIONS:
Overall Officials: Aldar Bourinbaiar, MD/PhD, Study Director — Immunitor LLC
Locations (1):
- Immunitor LLC, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at study completion

REFERENCES:
- See also: press release concerning preliminary results — http://www.prweb.com/releases/2014/06/prweb11965485.htm
- See also: Tarakanovskaya, M. G., Chinburen, J., Purevsuren, G., Munkhzaya, C., Batchuluun, P., Bat-Ireedui, P., … Bourinbaiar, A. S. (2015). Immunotherapy of liver cancer with hepcortespenlisimut-L: open-label Phase II clinical study in patients with advanced HCC. — http://doi.org/10.1186/2051-1426-3-S2-P200
- Available data/document: Abstract of 75-patient Phase II study: PMCID: PMC4649454 — http://doi.org/10.1186/2051-1426-3-S2-P200 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4649454/pdf/2051-1426-3-S2-P200.pdf